CLINICAL TRIAL: NCT05685121
Title: A Wearable Wrist-Worn Nerve Stimulator for Remediating Autonomic Dysfunction Associated With Persistent Post-Concussive Symptoms in Adolescents
Brief Title: A Wrist-Worn Nerve Stimulator for Remediating Persistent Post-Concussive Symptoms in Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of South Carolina (Other)
Collaborators: Prisma Health-Midlands (Other)
Responsible Party: Principal Investigator, Robert Davis Moore, Assistant Professor, University of South Carolina
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1926452
Record Dates: First submitted 2022-12-20; First posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Concussion, Brain
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apollo Neuro Group (Experimental): The group will use the Apollo Neuro device daily for six weeks as an adjunct to their standard treatment plan.
  Interventions: Device: Apollo Neuro
- Standard Treatment Group (No Intervention): The group will follow their standard treatment plan.

INTERVENTIONS:
Device: Apollo Neuro — The device is a wearable nerve stimulator.
  Arms: Apollo Neuro Group

SUMMARY:
The goal of this study is to test a wearable nerve stimulator in adolescents with persistent post-concussive symptoms. The main questions it aims to answer is whether the device will reduce clinical symptom burden, reduce cognitive deficits, and aid in the recovery of clinical symptoms.

Participants will wear the device daily for six weeks and complete a series of assessments.

DETAILED DESCRIPTION:
The primary aim of this study is to evaluate the effectiveness of the Apollo Neuro Device on remediating clinical symptoms, cognitive deficits and physical symptoms of those patients struggling with persisting post-concussive symptoms. The Apollo Neuro Device offers a convenient novel, non-invasive, non-habit-forming solution to improve performance and recovery under stress by delivering gentle wave-like vibrations to the body that improve autonomic nervous system balance in real time. The investigators will carry out a prospective study including any individual over the age of ten years presenting with persisting post-concussive symptoms. An Apollo Neuro Device will be offered as part of a treatment plan to patients with chronic neurological symptoms and will be used as an adjunct along with typical treatment. Patients will follow-up for a comprehensive evaluation, per discretion of specialty physicians and weekly symptom surveys will also be emailed to patients to track status. The results of this study will further the understanding of autonomic dysfunction symptomology and recovery and evaluate the effect of nerve stimulation as a means of mediating autonomic nervous system dysfunction in these patients.

ELIGIBILITY:
Inclusion Criteria:

* concussion diagnosis
* able to follow simple instruction
* able to sit upright in a chair for at least 30 minutes without rest

Exclusion Criteria:

* previous diagnosis of moderate or severe traumatic brain injury
* neuropsychiatric conditions of schizophrenia or bipolar disorder
* neurophysiological conditions of epilepsy, cerebral palsy, or severe sensory disorders

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-10-22 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Weekly changes in concussion symptoms | pre-intervention and weekly during the intervention
  Index of concussion symptoms using the Sport Concussion Assessment Tool 5 (SCAT-5). The SCAT-5 assesses the presence and severity of 22 common concussion symptoms, each rated on a scale from 0 (not present) to 6 (severe).
Changes in executive function | pre-intervention and after three and six weeks of device use
  Observed functioning will be reported by parents/guardians with the Behavior Rating Inventory of Executive Function (BRIEF). The BRIEF includes t-scores for comparison to sex- and age-normed data, with higher values indicating worse outcomes.
Change in concussion symptoms from pre-injury levels | pre-intervention and after three and six weeks of device use
  Current severity of concussion symptoms in comparison to severity prior to injury will be assessed with the Rivermead Post-Concussion Symptoms Questionnaire (RPQ). The RPQ includes 16 concussion symptoms that are rated in comparison to pre-injury levels from 0 to 4, with higher scores indicating more severe symptoms.
Changes in anxiety symptoms | pre-intervention and after three and six weeks of device use
  Intensity of anxiety symptoms assessed with the Beck Youth Inventory - Anxiety scale. Raw scores range from 0 to 60, with higher scores indicating more severe symptoms. T-scores are also included for comparison to normative data.
Changes in depression symptoms | pre-intervention and after three and six weeks of device use
  Index of depression symptoms using the Beck Youth Inventory - Depression scale. Raw scores range from 0 to 60, with higher scores indicating more severe symptoms. T-scores are also included for comparison to normative data.
Changes in psycho-affective health | pre-intervention and after three and six weeks of device use
  Index of psycho-affective health using the Profile of Mood States (POMS). Higher scores on the POMS indicate more intensely experienced mood states.
Changes in sleep disturbance | pre-intervention and after three and six weeks of device use
  Index of sleep disturbance using the Neurological Quality of Life (Neuro-QoL) sleep subscale. Raw scores range from 0 to 32, with higher scores indicating worse sleep disturbance. T-scores are also included for comparison to normative data.
Changes in pain severity | pre-intervention and after three and six weeks of device use
  Index of pain using the Neurological Quality of Life (Neuro-QoL) pain sub-scale. Raw scores range from 0 to 40, with higher scores indicating worse pain. T-scores are also included for comparison to normative data.
Changes in fatigue | pre-intervention and after three and six weeks of device use
  Index of pain using the Neurological Quality of Life (Neuro-QoL) fatigue sub-scale. Raw scores range from 0 to 32, with higher scores indicating worse fatigue. T-scores are also included for comparison to normative data.
Changes in headache burden | pre-intervention and after three and six weeks of device use
  Index of headache-related burden using the Headache Impact Test-6 (HIT-6). Scores range from 36-78 with higher scores indicating worse outcomes.
Changes in cognitive function | pre-intervention and after three and six weeks of device use
  Performance on the CogState, a validated brain injury cognitive battery.
Changes in vestibular/ocular motor screening | pre-intervention and after three and six weeks of device use
  Visuomotor processing issues associated with concussion, assessed via the Vestibular/Ocular Motor Screening assessment (VOMS).
Changes in balance | pre-intervention and after three and six weeks of device use
  Neuromuscular control assessed via the Modified Balance Error Scoring Screen (mBESS).
Changes in heart rate variability | pre-intervention and after three and six weeks of device use
  Cardio-autonomic function recorded at rest and while under increased physiological demand during a hand grip task.

CONTACTS AND LOCATIONS:
Locations (1):
- Prisma Health Pediatric Concussion Clinic, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No